CLINICAL TRIAL: NCT03707964
Title: Crisis Resource Management Improvement Through Intellectual Questioning of Authority
Acronym: CRITIQue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CRITIQue
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Medical Education, Simulation, Crisis Resource Management
Keywords: Medical Education; Simulation; Crisis Resource Management

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Deliberate deception (by not informing of the aim of assessing for ability to challenge authority) will be used to blind the participants. However, open disclosure and explanation of the rationale for deception will be conducted during the debriefing sessions and participants will be extensively counselled.
  The confederate specialist will also be blinded to the allocation of the control or intervention arm of participants.
  All sessions will be video recorded and assessed in random order by two independent raters blinded to group allocation, using the modified Advocacy-Inquiry Score (mAIS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Subjects allocated to the control arm will receive standard didactic interactive session on Advanced Cardiac Life Support (ACLS) principles, as part of their regular teaching schedule.
  Interventions: Other: Standard ACLS Training
- Intervention (Experimental): Subjects allocated to the intervention arm will receive education on crisis resource management (CRM) and teaching targeting the cognitive skills required to monitor and challenge a superior's decision, and conflict resolution tools, in addition to standard didactic interactive session on Advanced Cardiac Life Support (ACLS) principles.
  Interventions: Other: Crisis Resource Management Skill Training

INTERVENTIONS:
Other: Crisis Resource Management Skill Training — Focused crisis resource management training which targets at the cognitive skills needed to monitor and challenge a superior's decision.
  Arms: Intervention
Other: Standard ACLS Training — Standard didactic interactive session on Advanced Cardiac Life Support (ACLS) principles.
  Arms: Control

SUMMARY:
This is a randomized controlled trial examining the effectiveness of a teaching intervention on residents' and medical students' ability to challenge clearly wrong decisions by a superior during a simulated life-threatening crisis. Participants will be randomly allocated into the control or intervention arm. The intervention arm will receive education on crisis resource management (CRM) and teaching targeting the cognitive skills required to monitor and challenge a superior's decision, and conflict resolution tools. Participants will then take part in a simulation scenario 2 to 4 weeks later and will be assessed based on 6 challenge points, followed by a debrief session.

ELIGIBILITY:
Inclusion Criteria:

* Medical officers or Internal medicine, surgical and emergency medicine residents who are in their 2nd post-graduate year of training, or
* Phase V medical students from Yong Loo Lin School of Medicine, National University of Singapore

Exclusion Criteria:

* Refusal for informed consent, or
* Refusal for video recording during simulation sessions

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Effect of a teaching intervention on participants' ability to challenge clearly wrong decisions by a superior during a simulated life-threatening crisis | 20 minutes
  Comparison of the best modified Advocacy-Inquiry Score (mAIS) responses of the 6 challenge opportunities between the intervention and control groups. The mAIS is a modification of the Advocacy-Inquiry method which includes five scoring levels with the addition of a sixth level when a trainee attempts to take over management of the case.

SECONDARY OUTCOMES:
Influence of the confederate's gender on participant's ability to challenge incorrect decisions | 20 minutes
  Comparison of the median modified Advocacy-Inquiry Score (mAIS) responses between the subjects exposed to male versus female confederate specialist. The mAIS is a modification of the Advocacy-Inquiry method which includes five scoring levels with the addition of a sixth level when a trainee attempts to take over management of the case.

OTHER OUTCOMES:
Qualitative analysis of themes surrounding hierarchy and challenging authority | 10 minutes
  Themes elicited during open disclosure and discussion during debrief session with participants

CONTACTS AND LOCATIONS:
Overall Officials: Gene Chan, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No